CLINICAL TRIAL: NCT03105219
Title: IvaBradinE to Treat MicroalbumiNuria in Patients With Type 2 Diabetes and Coronary Heart Disease
Acronym: BENCH
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Shortfall in funding
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, Vice President, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFH20170403
Record Dates: First submitted 2017-04-03; First posted 2017-04-07 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Ivabradine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Urinary albumin excretion at 3 month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ivabradine (Experimental): Ivabradine 5mg twice a day (on day 0), heart rate evaluated at day 14 and 28 repeatedly, and the targeted value of heart rate 50-60bpm, the largest dosage 7.5mg twice a day.
  Interventions: Drug: Ivabradine
- Sham Comparator (Sham Comparator): Urinary albumin excretion (UAE) assessment will be performed before randomization (Day 0), 28-day after randomization (Day 28), and 90-day after randomization (Day 28).
  Interventions: Other: Sham Comparator

INTERVENTIONS:
Drug: Ivabradine — Ivabradine 5mg twice a day (on day 0), heart rate evaluated at day 14 and 28 repeatedly, and the targeted value of heart rate 50-60bpm, the largest dosage 7.5mg twice a day.
  Arms: Ivabradine
Other: Sham Comparator — Urinary albumin excretion (UAE) assessment will be performed before randomization (Day 0), 28-day after randomization (Day 28), and 90-day after randomization (Day 28).
  Arms: Sham Comparator

SUMMARY:
To explore the efficacy of Ivabradine for the treatment of microalbuminuria in patients with type 2 diabetes and coronary heart disease.

DETAILED DESCRIPTION:
This is a multi-center, randomized, open-label, investigator-initiated study with a parallel design. Patients with type 2 diabetes and coronary heart disease who are microalbuminuric [urinary albumin excretion (UAE): 30-500 mg/day], will be randomized after informed consent, in a 1:1 ratio to the following treatment groups: Group Α: Ivabradine 5mg twice a day (on day 0), heart rate evaluated at day 14 and 28 repeatedly, and the targeted value of heart rate 50-60bpm, the largest dosage 7.5mg twice a day.

Group Β: Placebo. Urinary albumin excretion (UAE) assessment will be performed before randomization (Day 0), 28-day after randomization (Day 28), and 90-day after randomization (Day 28).

ELIGIBILITY:
Inclusion Criteria:

* 1. Type 2 diabetes and coronary heart disease;
* 2. Urinary albumin excretion: 30-500mg/24h;
* 3. Sinus rhythm, and resting heart rate ≥ 70bpm;

Exclusion Criteria:

* 1. Renal dysfunction defined as eGFR < 30ml/min/1.73m^2;
* 2. Atrial flutter, and atrial fibrillation;
* 3. Resting heart rate < 70bpm;
* 4. Combined with non-dihydropyridine CCB;
* 5. UAE<30mg/24h, or > 500mg/24h;
* 6. Acute heart failure;
* 7. Low blood pressure (BP<90/50mmHg);
* 8. Acute myocardial infarction (<14 days);

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Urinary albumin excretion | 3 month
  Urinary albumin excretion at 3 month

SECONDARY OUTCOMES:
Serum creatinine | 3 month
  Serum creatinine at 3 month
Blood urea nitrogen | 3 month
  Blood urea nitrogen at 3 month
Cyscatin-c | 3 month
  Cyscatin-c at 3 month
Hypersensitive c-reactive protein (hsCRP) | 3 month
  Hypersensitive c-reactive protein (hsCRP) at 3 month
β2-microglobulin | 3 month
  β2-microglobulin at 3 month
Neutrophil gelatinase-associated lipocalin(NGAL) | 3 month
  Neutrophil gelatinase-associated lipocalin(NGAL) at 3 month
Albuminuria and urine creatinine ratio (ACR) | 3 month
  Albuminuria and urine creatinine ratio (ACR) at 3 month
N-acyl-β-D-glucosidase | 3 month
  N-acyl-β-D-glucosidase at 3 month
Retinol binding protein | 3 month
  Retinol binding protein at 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Shaoliang Chen, MD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No